CLINICAL TRIAL: NCT03838718
Title: REtroperitoneal SArcoma Registry (RESAR): Prospective Collection of Primary Retroperitoneal Sarcoma Patient's Data, Radiological and Pathological Material for the TransAtlantic Retroperitoneal Sarcoma Working Group
Brief Title: REtroperitoneal SArcoma Registry: an International Prospective Initiative
Acronym: RESAR
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: TransAtlantic Retroperitoneal Sarcoma Working Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: 201/16
Record Dates: First submitted 2018-03-29; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Retroperitoneal Sarcoma
Keywords: Sarcoma; Surgery; Multivisceral resection; Chemotherapy; Radiation Therapy; Patients' Registry
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Biopsies, Surgical specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgery is currently the only potentially curative treatment modality for localized retroperitoneal sarcoma (RPS). Available studies regarding oncologic outcomes are mainly retrospective in nature, and RPS are recognized as a rare disease. Therefore, prospective analysis of high quality data is a top priority.

Primary Objectives of this study are:

* to prospectively collect standardized clinical data and radiological and pathological material from primary RPS patients treated with surgery at reference centers.
* patient outcome will be evaluated in terms of overall survival (OS), disease-free survival (DFS), crude cumulative incidence (CCI) of local recurrence (LR) and distant metastasis (DM).

Secondary Objectives:

* to estimate the efficacy and safety of surgical treatment, including extended surgical approach to primary RPS;
* to prospectively evaluate the impact of multimodality therapy, including radiation therapy and chemotherapy;
* to identify clinical, radiological and pathological characteristics that may influence the oncological outcome or may be used as predictors of LR/DM/OS. These may be important biomarkers of disease;
* to utilize collected pathological material for research collaborations.

DETAILED DESCRIPTION:
Retroperitoneal sarcomas (RPS) are rare tumors accounting for 10-15% of all soft tissue sarcomas (STS). They arise between retroperitoneal organs and among vital structures (ie major abdominal vessels) in an anatomical compartment that is not readily accessible by physical examination. Four main histotypes account for about 80% of all cases: well-differentiated liposarcoma (WDLPS), dedifferentiated liposarcoma (DDLPS), leiomyosarcoma (LMS) and solitary fibrous tumor (SFT).

Compared to sarcomas at other anatomic sites, RPS are burdened by a higher local recurrence (LR) rate (50% at 5 years) and a poorer overall survival (OS) rate (50% at 5-years). The natural history of RPS as a whole group reflects the strong tendency of lipomatous tumors (WDLPS and DDLPS, which account for about 50% of RPS) to recur locally. Indeed, outcome of primary RPS is highly related to the histological subtype.

WDLPS are characterized by a relatively lower LR rate, negligible metastatic potential and a favorable overall survival. These tumors however, still may recur locally even years after the primary resection. Intermediate grade DDLPS are characterized by a strong tendency to recur locally and low metastatic potential. High grade DDLPS has a high risk of both local recurrence and distant metastasis. LMS are usually intermediate or high-grade tumors with a strong tendency to develop distant metastasis; with an adequate resection, it is relatively common to obtain a durable local control. Classic SFT usually fare well after surgery, with a low rate of local recurrence and distant metastasis.

Historically, surgery emerged as the only potentially curative option in the localized setting. In the last few years there has been lively debate as to how far should a surgeon resect in order to obtain a margin that could be considerate adequate. This issue is particularly challenging in this anatomical compartment where widening the surgical margins means resecting adjacent organs.

Since 2002 an 'extended' surgical approach has been proposed for primary RPS patients. The concept was that surgical margins could be improved by encompassing the tumor with en-bloc resection of adjacent organs. The aim was to obtain reduced local recurrence and improved survival. This approach has proven to be effective. In particular, this surgical approach has been supported by an experimental model, retrospective comparisons, pathology studies demonstrating adjacent organ involvement, and reports of high rates of residual tumor at re-excision after conventional (non-extended) primary surgery. Finally, this approach has been shown to be safe after both short and long term follow-up.

Radiotherapy is an option for RPS, especially in the preoperative setting, but currently the best evidence for efficacy comes form retrospective, mainly single-center, small size series. The results of such studies are controversial and high quality data are lacking. A randomized prospective study led by EORTC (STRASS) is ongoing but results are not expected for several years.

The role of chemotherapy in the localized disease is also still under investigation, especially in high grade tumors. So far, there is no agreement on the optimal treatment strategy, even within reference centers, regarding the use of both chemo- and radiotherapy. In the recent years European and North-American centers joined the panel of expert and this led to the formation of the TransAtlantic Retroperitoneal Sarcoma Working Group (TARPSWG), which now consists of more than 50 representatives from sarcoma centers from all over the world.

The aim of this collaboration is to expand the knowledge of the disease and formulate shared, standardized principles of treatment. A retrospective study has been carried out and recently published by the group to better define patients' outcome and prognostic factors after surgical resection of primary tumors. Other retrospective studies have been published focusing on post-relapse outcome, postsurgical morbidity and local recurrence treatment. This collaboration has also just recently led to the development of consensus guidelines for the treatment of primary and recurrent and metastatic RPS.

To take advantage of the group collaboration, TARPSWG promoted a prospective collection of clinical, radiological and pathologic data for RPS.

This study is aimed to prospectively collect standardized clinical data and radiological and pathological material from primary RPS patients treated with surgery at reference centers. Patient outcome will be evaluated in terms of overall survival (OS), disease-free survival (DFS), crude cumulative incidence (CCI) of local recurrence (LR) and distant metastasis (DM).

STUDY DESIGN

This is a prospective, multicentric observational study under the supervision of TARPSWG (TransAtlantic Retroperitoneal Sarcoma Working Group) aimed to prospectively collect clinical data and prospectively store radiological and pathological material from patients affected by primary RPS treated with surgery.

Patients with a diagnosis of primary RPS who meet the eligibility criteria will be invited to participate to the current study.

Eligible patients will receive full information on the type of surgery proposed and on the data and material (radiological and pathological) that will be collected. Eligible and informed patients who give their consent to participate will be included in the Prospective Cohort Study (PCS) and will be followed-up prospectively.

A data collection form including patient and tumor-related factors, treatment variables, follow-up findings, development of and time to local recurrence and status at follow-up has been constructed and shared among all the participating centers.

Each participating reference center will individually be able to have access to both cross sectional imaging (CT or MRI images) and pathological material (a representative formalin block of the tumor). Whenever possible patient identifiers will be removed and patient confidentiality will be maintained. Any data shared between institutions will be deidentified and all measures to conceal patient identifiers will be taken.

Each center will be responsible for data-entry and storage of its own patients' data, radiological examinations and pathological samples. At the time of the analysis each center is committed to provide the requested updated data to the group.

Follow-up will be based on clinical evaluation and on cross sectional imaging (CT scan of the thorax and abdomen and/or contrast enhanced MRI of the abdomen) every 4 months for the first 2 years, every 6 months until the 5th year and yearly thereafter.

The overall duration of the project has not been fixed.

Sample size

The number of patients we plan to include in this prospective multicenter study will be 400 patients per year.

STATISTICAL CONSIDERATIONS Continuous variables will be summarized with appropriate summary statistics such as the mean, median, standard deviation, minimum and maximum. Categorical variables will be tabulated with frequencies and percentages. We will evaluate OS, DFS, CCI of DM and LR and correlate this with clinicopathologic factors such as histology, grade, type of surgery, etc.

DATA COLLECTION Data entry will be performed by every participating center. Data will be collected in a standardized database, stored by every participating center, and shared with the group at the time of future studies. Data shared between institutions will be deidentified and whenever possible all measures to conceal patient identifiers and maintain patient confidentiality will be taken.

ETHICS It is the responsibility of the investigator to have prospective approval of the trial protocol, informed consent forms, and other relevant documents, from the IRB/IEC. All correspondence with the IRB/IEC should be retained in the Investigator File.

ELIGIBILITY:
Inclusion Criteria:

* primary RPS operated on in the participating center;
* age>18 years at the time of the first treatment (pediatric patients can not be included)
* histological confirmed diagnosis according to the WHO criteria done on biopsy or surgical specimen by dedicated sarcoma pathologist;
* radiological examinations performed (contrast enhanced abdominal CT scan and/or MRI) prior to surgical resection;
* signed informed consent form;
* adequate compliance of the patients to the plan of follow-up

Exclusion Criteria:

* age<18 years;
* recurrent tumor;
* benign retroperitoneal tumors;
* serious psychiatric disease that precludes informed consent or limits compliance;
* impossibility to ensure adequate follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a primary RPS amenable to surgical resection.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | 10 years
  Survival after surgery for primary RPS resection; any disease recurrence, local or distant, will be considered as an event at time of first radiological appearance.

SECONDARY OUTCOMES:
Overall Survival | 10 years
  Overall Survival computed from date of surgery
Crude cumulative incidence of Local recurrence | 10 years
  CCI of Local recurrence computed from date of surgery, and defined as intrabdominal recurrent disease after complete resection
Crude cumulative incidence of Distant metastasis | 10 years
  CCI of distant metastasis computed from date of surgery, and defined as hepatic recurrence and / or extrabdominal recurrent disease
Morbidity | 60 days
  Postsurgical morbidity according to Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Gronchi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Marco Fiore, MD, Study Director — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (22):
- United States (6):
  - University of Southern California (USC), Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory, Georgia
  - Brigham and Women's Hospital/Dana-Farber Cancer Institute, Boston, Massachusetts
  - The Ohio State University, Columbus, Ohio
- Peter MacCallum Cancer Center, Melbourne, Australia
- Canada (3):
  - Maisonneuve-Rosemont Hospital / University of Montreal, Montreal
  - The Ottawa Hospital, Ottawa
  - Mount Sinai / Princess Margaret, Toronto
- Institut Curie, Paris, France
- Germany (2):
  - University Medical Center and Medical Faculty Mannheim, University of Heidelberg, Mannheim
  - Ludwig Maximilian University, Munich
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Veneto Institute of Oncology, Padua
  - Ospedale Borgo Roma, Verona
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- Samsung Medical Center, Seoul, South Korea
- Hospital Clinico Universitario "Virgen de la Arrixaca", Murcia, Spain
- United Kingdom (2):
  - University Hospital Birmingham (Queen Elizabeth), Birmingham
  - Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gronchi A, Strauss DC, Miceli R, Bonvalot S, Swallow CJ, Hohenberger P, Van Coevorden F, Rutkowski P, Callegaro D, Hayes AJ, Honore C, Fairweather M, Cannell A, Jakob J, Haas RL, Szacht M, Fiore M, Casali PG, Pollock RE, Raut CP. Variability in Patterns of Recurrence After Resection of Primary Retroperitoneal Sarcoma (RPS): A Report on 1007 Patients From the Multi-institutional Collaborative RPS Working Group. Ann Surg. 2016 May;263(5):1002-9. doi: 10.1097/SLA.0000000000001447. PMID 26727100
- [Background] Trans-Atlantic RPS Working Group. Management of primary retroperitoneal sarcoma (RPS) in the adult: a consensus approach from the Trans-Atlantic RPS Working Group. Ann Surg Oncol. 2015 Jan;22(1):256-63. doi: 10.1245/s10434-014-3965-2. Epub 2014 Oct 15. PMID 25316486
- [Background] MacNeill AJ, Gronchi A, Miceli R, Bonvalot S, Swallow CJ, Hohenberger P, Van Coevorden F, Rutkowski P, Callegaro D, Hayes AJ, Honore C, Fairweather M, Cannell A, Jakob J, Haas RL, Szacht M, Fiore M, Casali PG, Pollock RE, Barretta F, Raut CP, Strauss DC. Postoperative Morbidity After Radical Resection of Primary Retroperitoneal Sarcoma: A Report From the Transatlantic RPS Working Group. Ann Surg. 2018 May;267(5):959-964. doi: 10.1097/SLA.0000000000002250. PMID 28394870
- [Derived] Benuzzi L, Iadecola S, Fiore M, Baia M, Colombo C, Radaelli S, Di Blasi E, Morosi C, Sanfilippo R, Callegaro D, Gronchi A. Pancreaticoduodenectomy and IVC resection in retroperitoneal sarcoma: Expanding the limits of feasible surgery. Eur J Surg Oncol. 2026 Jan;52(1):110547. doi: 10.1016/j.ejso.2025.110547. Epub 2025 Oct 26. PMID 41176815
- [Derived] Xiao M, Li X, Bu F, Ma S, Yang X, Chen J, Zhao Y, Cananzi F, Luo C, Min L. Molecular feature-based classification of retroperitoneal liposarcoma: a prospective cohort study. Elife. 2025 May 23;14:RP100887. doi: 10.7554/eLife.100887. PMID 40407808
- [Derived] Zhao Y, Qin D, Li X, Wang T, Zhang T, Rao X, Min L, Wan Z, Luo C, Xiao M. Identification of NINJ1 as a novel prognostic predictor for retroperitoneal liposarcoma. Discov Oncol. 2024 May 11;15(1):155. doi: 10.1007/s12672-024-01016-x. PMID 38733554
- See also: website of Trans-Atlantic Retroperitoneal Sarcoma Working Group — http://www.tarpswg.org